CLINICAL TRIAL: NCT03372330
Title: Prevalence and Outcomes of Peripheral Artery Disease in Sepsis Patients in the Medical Intensive Care Unit
Brief Title: Peripheral Artery Disease and Sepsis Outcomes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Other Study IDs: 106-044-E
Record Dates: First submitted 2017-12-10; First posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Peripheral Artery Disease; Peripheral Artery Occlusion; Sepsis; Diagnosis
Keywords: peripheral artery disease; sepsis
MeSH Terms: conditions — Peripheral Arterial Disease; Sepsis; Disease | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis with PAD: Patients admitted to the intensive care unit with the diagnosis of sepsis (quick SOFA score >=2) and with ankle-brachial index < 0.9 or vascular Duplex confirmed peripheral artery disease.
  * Standard care for sepsis and PAD
  Interventions: Drug: Standard care for sepsis and PAD
- Sepsis without PAD: Patients admitted to the intensive care unit with the diagnosis of sepsis (quick SOFA score >=2) and with ankle-brachial index >= 0.9 or vascular Duplex found no evidence of peripheral artery disease.
  * Standard care for sepsis
  Interventions: Drug: Standard care for sepsis

INTERVENTIONS:
Drug: Standard care for sepsis and PAD — The standard medications care for the patient with PAD included antiplatelet agents.
  Other Names: Sepsis with PAD
  Groups: Sepsis with PAD
Drug: Standard care for sepsis — The standard care for the patient with sepsis.
  Other Names: Sepsis without PAD
  Groups: Sepsis without PAD

SUMMARY:
The peripheral artery disease (PAD) prevalence is high in the elderly, the diabetic patients, and the patients receiving hemodialysis. To date, there is no guideline recommendation on the screening of PAD in patients admitted to the medical intensive care unit (MICU) for sepsis.

We conducted a prospective cohort study focusing on patients admitted to the MICU with the main diagnosis of sepsis. The ankle-brachial indexes are performed within 24 hours after admission. Invasive arterial line monitoring and standard non-invasive measurements are collected. After confirmation of PAD, standard anti-platelet treatments (aspirin and cilostazol) are initiated. The survival before and after the conduction of this trial is compared to historical records. The outcomes including all-cause mortality, stroke, myocardial infarction, minor amputation, major amputation, and prolonged ventilator dependent are to be collected.

DETAILED DESCRIPTION:
This is a prospective observational study focusing on peripheral artery disease (PAD) in patients admitting to intensive care units with a diagnosis of sepsis. The sepsis is defined by the quick SOFA score. The primary outcome is all-cause mortality. The secondary outcomes included stroke, myocardial infarction, amputation, and prolonged mechanical ventilation.

We plan to enroll 150 patients. Patients will be grouped into patients with PAD and patients without PAD. We then compare them in the following parameters: clinical data, laboratory data, survival and other outcome data. Two-sample student's t-tests will be used for the comparisons of continuous variables. Chi-square test will be used to detect the difference between categorical variables. The difference is considered statistically significant if P < 0.05. All statistics works were analyzed using the SPSS 17.0 software (Chicago, IL, USA), R software (Gimc packages).

ELIGIBILITY:
Inclusion Criteria:

* sepsis patients admitted to the MICU meeting quick SOFA score >= 2 points

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the medical intensive care units meeting sepsis definition.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-09-11 (Actual); Primary Completion 2018-09-10 (Estimated); Study Completion 2019-09-10 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality at 30-day | 30 days
  All-cause mortality at 30 days

SECONDARY OUTCOMES:
Myocardial infarction | 30 days
  Myocardial infarction at 30 days
Stroke | 30 days
  Ischemic stroke at 30 days
Amputation | 30 days
  Amputation, either major or minor at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Mu-Yang Hsieh, MD, Principal Investigator — National Taiwan University Hospital Hsin-Chu Branch
Locations (1):
- National Taiwan University Hospital, Hsin-Chu Branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tseng H, Liao MT, Keng LT, Chang CH, Zeng YZ, Hsieh MY. Impact of Abnormal Ankle Brachial Index on Sepsis Survival: One-Year Prospective Study Results. Acta Cardiol Sin. 2024 Sep;40(5):627-634. doi: 10.6515/ACS.202409_40(5).20240528A. PMID 39308652

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/30/NCT03372330/Prot_SAP_000.pdf